CLINICAL TRIAL: NCT06577714
Title: Ablation Guided Via Precision Imaging Using Electromechanical Wave Imaging
Acronym: AGAPE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Elaine Y. Wan, Associate Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAU7964
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the data manager and biostatistician will retain the master list that identifies the randomization allocation and be unblinded. The Data Safety and Monitoring Board and all those who contact patients, the steering PIs, and advisory committee will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- 3D EWI (Active Comparator): Electromechanical Wave Imaging (EWI) is an ultrasound-based technique that takes 10-15 minute to non-invasively image arrhythmias by visualizing the electromechanical wave corresponding to electromechanical coupling. A full 3D EWI noninvasive ultrasound technique which can construct an entire 4 chamber cardiac activation map using a single heartbeat of arrhythmia acquired in one apical transthoracic echocardiographic image.
  Interventions: Diagnostic Test: Electromechanical wave imaging (EWI)
- Standard of Care (No Intervention): Ablation without image guided ablation

INTERVENTIONS:
Diagnostic Test: Electromechanical wave imaging (EWI) — EWI is a high-frame rate ultrasound technique that images the electromechanical wave corresponding to the propagation of the onset of myocardial contraction in response to electrical activation, namely electromechanical coupling.
  Arms: 3D EWI

SUMMARY:
Atrial and ventricular cardiac arrhythmias are serious public health problems in the United States, affecting over 5% of Americans and are major causes of stroke and heart failure leading to increased morbidity and mortality. This proposed clinical trial will determine how electromechanical wave imaging (EWI), a non-invasive ultrasound precision imaging modality, can effectively diagnose and determine the mechanism of the arrhythmia and impact personalized treatment of cardiac arrhythmias. Participants who are already scheduled for electrophysiology study will receive EWI prior to their study. Half of participants will randomly have their EWI imaging data available for their electrophysiologist to analyze and potentially affect procedure planning and execution. Across all participants the results of EWI and the electrophysiology study will be compared to determine EWI accuracy at diagnosing arrhythmias. Participants whose electrophysiologists had access to EWI data will be compared against those without access to determine if EWI data led to improved procedure efficiency and outcomes.

DETAILED DESCRIPTION:
Cardiac arrhythmias are a major cause of morbidity and mortality affecting over 5% of Americans. Arrhythmias have become increasingly prevalent due to an aging population with diabetes, heart failure and hypertension, which has led to an increasing number of invasive electrophysiology studies and catheter ablations. Understanding of the cardiac arrhythmia mechanism, if it is focal or reentrant, and the specific location of the arrhythmia origin is limited by the current first-line, standard of care, noninvasive diagnostic test - the 12-lead electrocardiogram (ECG), which is dependent on physician subjective interpretation. Furthermore, it does not present the arrhythmia in an easily visualized, three-dimensional, anatomical manner for patients or physicians to understand. Other noninvasive mapping techniques such as ECG imaging (ECGI) or virtual-heart technology, requires additional preprocedural imaging such as computed tomography which exposes patient to radiation, or magnetic resonance imaging which is costly. Over ten years, the collaborative team effort between Cardiac Electrophysiology and Biomedical Engineering at Columbia University Irving Medical Center, has developed Electromechanical Wave Imaging (EWI), an ultrasound-based technique that takes 10-15 minutes to non-invasively image arrhythmias by visualizing the electromechanical wave corresponding to electromechanical coupling. A new technique, a full 3D EWI noninvasive ultrasound technique, has been developed which can construct an entire 4 chamber cardiac activation map using a single heartbeat of arrhythmia acquired in one apical transthoracic echocardiographic image. This study involves three aims which will validate non-invasive 3D EWI to high density activation maps (HDAM) acquired during invasive electrophysiology study and demonstrate its clinical impact to shorten procedural times and improve clinical outcomes in a randomized clinical trial. The investigators will study patients with manifest pre-excitation such as Wolff-Parkinson-White syndrome, atrial tachycardia, atrial flutter, premature atrial complexes, premature ventricular complexes and ventricular tachycardia. This study aims to demonstrate that 3D EWI is an invaluable tool for pre-ablation planning to (1) provide target localization, (2) diagnose the mechanism of the arrhythmia, as focal or macro-reentrant arrhythmia, useful in decision-making for systemic anticoagulation and (3) improve ablation outcomes in terms of mapping/procedure times and number of ablation lesions.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years of age
* Able to give consent for the study
* Scheduled for Invasive Electrophysiology Study (EPS) +/- ablation for atrial tachycardia (AT), atrial flutter (AFL), Wolff-Parkinson-White syndrome (WPW) or premature atrial complexes/premature ventricular complexes (PAC/PVCs)

Exclusion Criteria:

* Patient is not in clinical arrhythmia at the time of scan despite leg lifts, or intravenous isoproterenol/dobutamine infusion
* Patient is not able to comply with study protocol due to cognitive impairment, severe mental illness, or planned moved during the study period
* Treating physician does not agree with enrollment
* Patient does not speak English or Spanish
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Proportions of correct predictions for location of arrhythmia in both standard of care ECG reads compared to EWI maps | Up to 1 week
  A correct prediction is defined as if it correctly identifies the location of the arrhythmia. A correct prediction is defined as if it correctly identifies the location of the arrhythmia. The 3D EWI maps will be generated prior to procedure and acquisition of the image takes usually takes 15 minutes. Data processing will take at least 1-3 days and will be available prior to the start of the electrophysiology study. Comparative analysis of the results from 3D EWI to the 3D high density electroanatomical maps will take place up to 1 week after the procedure to compare the prediction of target ablation to the area of ablation success.
Proportions of correct predictions for mechanism of arrhythmia in both standard of care ECG reads compared to EWI maps | Up to 1 week
  A correct prediction is defined as 1) a method correctly identifies an arrhythmia as focal or macro-reentrant The 3D EWI maps will be generated prior to procedure and acquisition of the image takes usually takes 15 minutes. Data processing will take at least 1-3 days and will be available prior to the start of the electrophysiology study. Comparative analysis of the results from 3D EWI to the 3D high density electroanatomical maps will take place up to 1 week after the procedure to compare the predicted mechanism to the invasively acquired activation map revealing the true mechanism of the arrhythmia

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No